CLINICAL TRIAL: NCT05020314
Title: Healthy Weight Clinic: Packaging and Spreading Proven Pediatric Weight Management Interventions for Use by Low-Income Families, Childhood Obesity Research Demonstration Project (CORD) 3.0
Brief Title: Pediatric Healthy Weight Clinic
Acronym: CORD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); American Academy of Pediatrics (Other)
Responsible Party: Principal Investigator, Lauren G. Fiechtner, M.D., Director of Nutrition, Division of Gastroenterology and Pediatric Health Outcomes Research, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021P000258; 2023P003302
Record Dates: First submitted 2021-08-12; First posted 2021-08-25 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Children receiving care at the implementation sites, and who are referred to and attend the Healthy Weight Clinic will receive the intervention as described.
  A sample of demographically matched children who did not receive the intervention will serve as a comparison group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinically Based: Healthy Weight Clinic (Experimental)
  Interventions: Behavioral: Healthy Weight Clinic

INTERVENTIONS:
Behavioral: Healthy Weight Clinic — Patients meet with a multi-disciplinary team over a 12 month period. In addition to the clinical visits, group visits, and phone calls, patients will also receive education materials, community resources, and an optional text messaging/social media library of messages.

SUMMARY:
The overall goal of this study is to increase access to and adoption of the Healthy Weight Clinic package in primary care settings serving low income families in the United States who have a disproportionately high prevalence of childhood obesity. Two federally-qualified health centers in Mississippi and two health centers in Massachusetts will be implementing a Healthy Weight Clinic Program. The Healthy Weight Clinic is staffed by a medical provider, a Dietitian/Nutritionist, and a Community Healthy Worker. Patients attend individual medical visits (once per month for 12 months) with the multidisciplinary team, group visits led by a member of the team (once per month for 6 months), and phone follow-up between visits. All patients who receive care at the pilot implementation sites will be exposed to the systems-level intervention. A subset of patients will be invited to participate in a research evaluation of the program.

ELIGIBILITY:
Inclusion Criteria:

* child is age 2 through 18 years at referral
* child's BMI meets or exceeds the 85th percentile for age and sex
* parent can read and respond to interviews and questionnaires in English or Spanish
* received care at one of the participating pilot sites

Exclusion Criteria:

* children who do not have at least one parent who can report on their child's daily activities for 1 year
* families who plan to leave their pediatric health center in the next year
* children who have conditions or take medications that substantially interfere with growth, physical activity, or dietary recommendations

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 191 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Child BMI at 12 months | 0-12 months
  Weight and height will be combined to report BMI in kg/m^2 based on CDC growth curves.
Change in Child BMI percent of the 95th percentile at 12 months | 0-12 months
  Weight and height will be combined to report BMI in kg/m^2 based on CDC growth curves.
Change in Child BMI z-score at 12 months | 0-12 months
  Weight and height will be combined to report BMI z-score based on CDC growth curves

SECONDARY OUTCOMES:
Change in Child Quality of Life at 12 months based on Sizing Them Up Questionnaire | 0-12 months
Change in Child Binge Eating at 12 months based on Questionnaire | 0-12 months
Change in Child Parental Stress at 12 months based on Questionnaire | 0-12 months
Change in Family Food Insecurity at 12 months based on Hunger Vital Signs Questionnaire | 0-12 months
Change in Child Nutrition at 12 months based on Questionnaire | 0-12 months
Change in Child Physical Activity at 12 months based on Questionnaire | 0-12 months
Change in Child Sleep at 12 months based on Questionnaire | 0-12 months
Change in Child Screen Time at 12 months based on Questionnaire | 0-12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual-level data may be shared upon request, under the conditions that an analysis plan is prepared and approved by the PI/Co-Is, IRB approval has been obtained, and all necessary data sharing agreements have been executed.
Supporting Information: Study Protocol, ICF
Time Frame: Data can be requested by emailing the PI or Project Manager.
Access Criteria: 1. An analysis plan is prepared and approved by the PI/Co-Is,
  2. IRB approval has been obtained, and
  3. All necessary data sharing agreements have been executed.

REFERENCES:
- [Background] Fiechtner L, Sierra Velez D, Ayala SG, Castro I, Lindros J, Perkins M, Baker A, Salmon J, Biggs V, Cannon-Smith G, Smith JD, Simione M, Gortmaker SL, Taveras EM. Planned Evaluation of the Healthy Weight Clinic Pediatric Weight Management and Implementation: Massachusetts-CORD 3.0. Child Obes. 2021 Sep;17(S1):S55-S61. doi: 10.1089/chi.2021.0178. PMID 34569842
- [Background] Fiechtner L, Castro I, Ayala SG, Velez DS, Lindros J, Perkins M, Baker A, Salmon J, Biggs V, Cannon-Smith G, Smith JD, Simione M, Gortmaker SL, Taveras EM. Design and Approach of the Healthy Weight Clinic Pediatric Weight Management Intervention Package and Implementation: Massachusetts-CORD 3.0. Child Obes. 2021 Sep;17(S1):S48-S54. doi: 10.1089/chi.2021.0177. PMID 34569841
- [Background] Sierra-Velez D, Gundewar A, Persaud A, Simione M, Castro I, Perkins M, Lindros J, Salmon J, Smith JD, Taveras EM, Fiechtner L. Stakeholders' perception of factors influencing adoption of a pediatric weight management intervention: a qualitative study. Front Public Health. 2023 Oct 13;11:1045618. doi: 10.3389/fpubh.2023.1045618. eCollection 2023. PMID 37900042